CLINICAL TRIAL: NCT07196722
Title: A Phase 2b/3 Randomized, Double-blind, Placebo-Controlled, Parallel Group, Multicenter Protocol to Evaluate the Efficacy and Safety of Icotrokinra in Participants With Moderately to Severely Active Crohn's Disease
Brief Title: A Study of Icotrokinra in Participants With Moderately to Severely Active Crohn's Disease
Acronym: ICONIC-CD
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 77242113CRD3001; 77242113CRD3001 (Other: Janssen Research & Development, LLC); 2025-521382-27-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2025-09-22; First posted 2025-09-29 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Induction Study 1: Icotrokinra Dose 1 (Experimental): Participants will receive Icotrokinra dose 1 in Induction Study 1 up to Week 12. Subsequent treatment will be determined by the participant's response status at Week 12.
  Interventions: Drug: Icotrokinra
- Induction Study 1: Icotrokinra Dose 2 (Experimental): Participants will receive Icotrokinra dose 2 in Induction Study 1 up to Week 12. Subsequent treatment will be determined by the participant's response status at Week 12.
  Interventions: Drug: Icotrokinra
- Induction Study 1: Placebo (Placebo Comparator): Participants will receive matching placebo in Induction Study 1 up to Week 12. Subsequent treatment will be determined by the participant's response status at Week 12.
  Interventions: Drug: Placebo
- Induction Study 2: Icotrokinra (Experimental): Participants will receive Icotrokinra at the dose regimen determined in Induction Study 1 up to Week 12. Subsequent study treatment will be determined by the participant's response status at Week 12.
  Interventions: Drug: Icotrokinra
- Induction Study 2: Placebo (Placebo Comparator): Participants will receive matching placebo for up to Week 12. Subsequent study treatment will be determined by the participant's response status at Week 12.
  Interventions: Drug: Placebo
- Maintenance Study: Icotrokinra Dose 1 (Experimental): Participants who were receiving icotrokinra in either induction studies 1 or 2 and were in response at Week 12 of the induction study will be randomized to receive icotrokinra maintenance dose 1. Participants receiving Icotrokinra Dose 1 and meeting criteria for loss of response during the Maintenance Study will be eligibile for a single blinded dose adjustment to Icotrokinra Dose 2. After completion of the Maintenance Study through Week 40, eligible participants can participate in long-term extension (LTE).
  Interventions: Drug: Icotrokinra
- Maintenance Study: Icotrokinra Dose 2 (Experimental): Participants who were receiving icotrokinra in either induction studies 1 or 2 and were in response at Week 12 of the induction study will be randomized to receive icotrokinra maintenance dose 2. Participants who were non-responders at Week 12 of the induction studies will also receive icotrokinra maintenance dose 2 but will not be randomized. After completion of the Maintenance Study through Week 40, eligible participants can participate in LTE.
  Interventions: Drug: Icotrokinra
- Maintenance Study: Placebo (Placebo Comparator): Participants who were receiving icotrokinra in either induction studies 1 or 2 and were in response at Week 12 will be randomized to receive placebo. Participants receiving placebo in induction studies 1 or 2 and in response at Week 12 of the induction study will continue to receive placebo during maintenance on non-randomized basis. Placebo non-responders from induction study will receive icotrokinra maintenance dose 2 on a non-randomized basis and will be assessed for response at Week 12.
  Participants receiving placebo and meeting criteria for loss of response during the Maintenance Study will be eligible for a single blinded dose adjustment to icotrokinra dose 2. After completion of the Maintenance Study through Week 40, eligible participants can participate in LTE.
  Interventions: Drug: Icotrokinra; Drug: Placebo

INTERVENTIONS:
Drug: Icotrokinra — Icotrokinra will be administered orally, daily.
  Other Names: JNJ-77242113
  Arms: Induction Study 1: Icotrokinra Dose 1; Induction Study 1: Icotrokinra Dose 2; Induction Study 2: Icotrokinra; Maintenance Study: Icotrokinra Dose 1; Maintenance Study: Icotrokinra Dose 2; Maintenance Study: Placebo
Drug: Placebo — Matching placebo will be administered orally, daily.
  Arms: Induction Study 1: Placebo; Induction Study 2: Placebo; Maintenance Study: Placebo

SUMMARY:
The purpose of this study is to evaluate how-well icotrokinra works (clinical efficacy) and how safe it is (safety) in participants with moderately to severely active Crohn's disease (CD; a long-term condition causing severe inflammation of the intestinal tract).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CD established at least 12 weeks before screening including both endoscopic evidence and a histopathology report consistent with a diagnosis of CD
* Moderately to severely active CD based on CDAI criteria, defined as baseline (Week I-0) CDAI score >=220 but <=450 and either mean daily SF count >=4, or mean daily AP score >=2
* Moderately to severely active CD based on SES-CD criteria assessed by baseline (Week I-0) endoscopic evidence of active ileal and/or colonic CD as assessed during central review of the screening video ileocolonoscopy defined as a SES-CD >= 6 for participants with colonic or ileocolonic disease, and SES-CD >= 4 for participants with isolated ileal disease, based on the presence of ulceration in any 1 of the 5 ileocolonic segments
* A female participant of childbearing potential must have a negative highly sensitive serum pregnancy test (beta-hCG) at screening and a negative urine pregnancy test at Week I-0 prior to administration of study intervention and agree to further pregnancy tests
* Demonstrated an inadequate response, loss of response, or failure to tolerate previous conventional therapy (advanced drug therapy [ADT]-naïve) or advanced therapy defined as biologics and/or advanced oral agents for the treatment of CD (ADT-inadequate responder [IR]) as defined in the protocol

Exclusion criteria:

* Has complications of CD, such as symptomatic strictures or stenoses, short gut syndrome, or any other manifestation, that may require surgery while enrolled in the study and/or could impair the use of instruments (such as CDAI) to assess response to study intervention
* Presence of a stoma or ostomy
* Participants with presence of active fistulas may be included if there is no surgery needed
* Colonic resection within 24 weeks before baseline or any other major surgery performed within 12 weeks before baseline
* Presence on screening colonoscopy of adenomatous colon polyps outside of an area of known colitis not removed before randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1092 (Estimated)
Dates: Start 2025-10-03 (Actual); Primary Completion 2028-09-19 (Estimated); Study Completion 2032-10-06 (Estimated)

PRIMARY OUTCOMES:
Induction Study 1: Number of Participants with Clinical Response at Week 12 | At Week 12
  Clinical response is defined as a greater than or equal to (>=) 100-point reduction from baseline in Crohn's Disease Activity Index (CDAI) score. CDAI scores range from 0 to approximately 600. Higher score indicates higher disease activity.
Induction Study 2: Number of Participants with Clinical Remission at Week 12 (Co-Primary Endpoint) | At Week 12
  Clinical remission is defined as CDAI score less than (<) 150. CDAI scores range from 0 to approximately 600. Higher score indicates higher disease activity.
Induction Study 2: Number of Participants with Endoscopic Response at Week 12 (Co-Primary Endpoint) | At Week 12
  Endoscopic response is defined as greater than (>) 50% improvement from baseline in Simple Endoscopic Score for Crohn's Disease (SES-CD) score or a decrease of at least 2 points in participants with a baseline score of 4 and isolated ileal disease. SES-CD score can range from 0 to 56. Higher scores indicating more severe disease.
Maintenance Study: Number of Participants with Clinical Remission at Week 40 (Co-Primary Endpoint) | At Week 40
  Clinical remission is defined as CDAI score < 150. CDAI scores range from 0 to approximately 600. Higher score indicates higher disease activity.
Maintenance Study: Number of Participants with Endoscopic Response at Week 40 (Co-Primary Endpoint) | At Week 40
  Endoscopic response is defined as > 50% improvement from baseline in SES-CD score or a decrease of at least 2 points in participants with a baseline score of 4 and isolated ileal disease. SES-CD score can range from 0 to 56. Higher scores indicating more severe disease.

SECONDARY OUTCOMES:
Induction Study 1: Number of Participants with Clinical Remission at Week 12 | At Week 12
  Clinical remission is defined as CDAI score < 150. CDAI scores ranging from 0 to approximately 600. Higher score indicates higher disease activity.
Induction Study 1: Number of Participants with Endoscopic Response at Week 12 | At Week 12
  Endoscopic response is defined as > 50% improvement from baseline in SES-CD score or a decrease of at least 2 points in participants with a baseline score of 4 and isolated ileal disease. SES-CD score can range from 0 to 56. Higher scores indicating more severe disease.
Induction Study 1: Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 4 weeks after last dose of study drug (i.e., up to Week 16)
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product that does not necessarily have a causal relationship with the intervention. An SAE is any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product and is medically important.
Induction Study 2: Number of Participants with Patient Reported Outcomes (PRO)-2 Remission at Week 12 | At Week 12
  PRO-2 remission is defined as an abdominal pain (AP) mean daily score less than or equal to (<=) 1 and stool frequency (SF) mean daily score <= 2.8, and no worsening of AP or SF from baseline.
Induction Study 2: Number of Participants with Clinical Response at Week 12 | At Week 12
  Clinical response is defined as a >= 100-point reduction from baseline in CDAI score.
Induction Study 2: Number of Participants Reporting Both Clinical Remission and Endoscopic Response at Week 12 | At Week 12
  Clinical remission is defined as CDAI score < 150. Endoscopic response is defined as > 50% improvement from baseline in SES-CD score or a decrease of at least 2 points in participants with a baseline score of 4 and isolated ileal disease. This is a composite endpoint defined to measure achievement of both clinical remission and endoscopic response at the participant level.
Induction Study 2: Number of Participants with Clinical Response at Week 4 | At Week 4
  Clinical response is defined as a >= 100-point reduction from baseline in CDAI score.
Induction Study 2: Number of Participants with Endoscopic Remission at Week 12 | At Week 12
  Endoscopic remission is defined as SES-CD <= 4 with at least a 2-point reduction from baseline and no sub score >1 in any individual component.
Induction Study 2: Number of Participants with Deep Remission at Week 12 | At Week 12
  Deep remission is a composite endpoint defined as achieving both clinical remission and endoscopic remission at the participant level. Clinical remission is defined as CDAI score < 150-point. Endoscopic remission is defined as SES-CD <= 4 with at least a 2-point reduction from baseline and no sub score >1 in any individual component.
Induction Study 2: Number of Participants with Inflammatory Bowel Disease Questionnaire (IBDQ) Remission at Week 12 | At Week 12
  IBDQ remission is defined as IBDQ score >= 170. IBDQ is a validated, 32-item, self-reported questionnaire for participants with inflammatory bowel disease (IBD) that will be used to evaluate the disease-specific health-related quality of life (HRQoL) across 4 dimensional scores: bowel symptoms (loose stools, abdominal pain), systemic symptoms (fatigue, altered sleep pattern), social function (work attendance, need to cancel social events), and emotional function (anger, depression, irritability). Scores range from 32 to 224, with higher scores indicating better outcomes.
Induction Study 2: Number of Participants with Fatigue Response at Week 12 | At Week 12
  Fatigue response is defined as a >= 7 point reduction in the patient reported outcomes measurement information system (PROMIS)-Fatigue Short Form 7a total score from baseline. The PROMIS fatigue SF-7a contains 7 items evaluating fatigue-related symptoms (that is, tiredness, exhaustion, mental tiredness, and lack of energy) and associated impacts on daily activities (that is, activity limitations related to work, self-care, and exercise). Item responses are rated on a five-point scale ranging from "never" to "always". Higher scores indicate more fatigue.
Induction Study 2: Number of Participants with Clinical Remission at Week 4 | At Week 4
  Clinical remission is defined as CDAI score< 150.
Induction Study 2: Number of Participants with AEs and SAEs | Up to 4 weeks after last dose of study drug (i.e., up to Week 16)
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product that does not necessarily have a causal relationship with the intervention. An SAE is any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product and is medically important.
Maintenance Study: Number of Participants with PRO-2 remission at Week 40 | At Week 40
  PRO-2 remission is defined as an abdominal pain (AP) mean daily score <= 1 and stool frequency (SF) mean daily score <= 2.8, and no worsening of AP or SF from baseline.
Maintenance Study: Number of Participants with Endoscopic Remission at Week 40 | At Week 40
  Endoscopic remission is defined as SES-CD <= 4 with at least a 2-point reduction from baseline and no sub score >1 in any individual component.
Maintenance Study: Number of Participants with 90-Day Corticosteroid-Free Clinical Remission at Week 40 | At Week 40
  90-day corticosteroid-free clinical remission is defined as the clinical remission at the visit and not receiving corticosteroids for 90 days prior to the visit. Clinical remission is defined as CDAI score < 150.
Maintenance Study: Number of Participants with Maintenance of Clinical Remission at Week 40 | At Week 40
  Participants with clinical remission at Week 40 among those with clinical remission at Week 0 of the maintenance study will be analyzed. Clinical remission is defined as CDAI score < 150.
Maintenance Study: Number of Participants Reporting Both Clinical Remission and Endoscopic Response at Week 40 | At Week 40
  Clinical remission is defined as CDAI score < 150. Endoscopic response is defined as > 50% improvement from baseline in SES-CD score or a decrease of at least 2 points in participants with a baseline score of 4 and isolated ileal disease. This is a composite endpoint defined to measure achievement of both clinical remission and endoscopic response at the participant level.
Maintenance Study: Number of Participants with Deep Remission at Week 40 | At Week 40
  Deep remission is a composite endpoint defined as achieving both clinical remission and endoscopic remission at the participant level. Clinical remission is defined as CDAI score < 150. Endoscopic remission is defined as SES-CD <= 4 with at least a 2-point reduction from baseline and no sub score >1 in any individual component.
Maintenance Study: Number of Participants with IBDQ Remission at Week 40 | At Week 40
  IBDQ remission is defined as IBDQ score >= 170. IBDQ is a validated, 32-item, self-reported questionnaire for participants with IBD that will be used to evaluate the disease-specific HRQoL across 4 dimensional scores: bowel symptoms (loose stools, abdominal pain), systemic symptoms (fatigue, altered sleep pattern), social function (work attendance, need to cancel social events), and emotional function (anger, depression, irritability). Scores range from 32 to 224, with higher scores indicating better outcomes.
Maintenance Study: Number of Participants with Fatigue Response at Week 40 | At Week 40
  Fatigue response is defined as a >= 7 point reduction in the PROMIS-Fatigue Short Form 7a total score from baseline. The PROMIS fatigue SF-7a contains 7 items evaluating fatigue-related symptoms (that is, tiredness, exhaustion, mental tiredness, and lack of energy) and associated impacts on daily activities (that is, activity limitations related to work, self-care, and exercise). Item responses are rated on a five-point scale ranging from "never" to "always". Higher scores indicate more fatigue.
Maintenance Study : Number of Participants with AEs and SAEs | Up to 4 weeks after last dose of study drug (i.e., up to Week 44)
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product that does not necessarily have a causal relationship with the intervention. An SAE is any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product and is medically important.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (181):
- United States (37):
  - AZ Gastro Care, Chandler, Arizona
  - Clinnova Research, Anaheim, California
  - Alliance Research Institute, LLC - Canoga Park, Canoga Park, California
  - Southern California Research Center, Coronado, California
  - Om Research LLC, Lancaster, California
  - TLC Clinical Research Inc, Los Angeles, California
  - GastroIntestinal Bioscience, Los Angeles, California
  - Om Research LLC, Oxnard, California
  - Clinical Applications Laboratories, Inc, San Diego, California
  - Medical Associates Research Group, Inc., San Diego, California
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Nuvance Health Danbury Hospital, Danbury, Connecticut
  - American Institute of Research, Cutler Bay, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - Green Leaf Clinical Trials, Jacksonville, Florida
  - Florida Research Center Inc., Lakewood Rch, Florida
  - Sanchez Clinical Research, Inc, Miami, Florida
  - GCP Clinical Research, Tampa, Florida
  - Children's Center for Digestive Health Care, Atlanta, Georgia
  - Gastroenterolgy Associates of Central GA, Macon, Georgia
  - Kansas Gastroenterology, LLC, Wichita, Kansas
  - Tri-State Gastroenterology Assoc, Crestview Hills, Kentucky
  - Gastroenterology Clinic of Acadiana, Lafayette, Louisiana
  - Delta Research Partners, LLC, West Monroe, Louisiana
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Westchester Putnam Gastroenterology, Carmel, New York
  - Manhattan Clinical Research LLC, New York, New York
  - New York Gastroenterology Associates, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Gastro Intestinal Research Institute of Northern Ohio LLC, Westlake, Ohio
  - Digestive Disease Specialists Inc, Oklahoma City, Oklahoma
  - The Oregon Clinic, Portland, Oregon
  - Susquehanna Research Group, Harrisburg, Pennsylvania
  - Digestive Disease Associates, Rock Hill, South Carolina
  - DFW Clinical Trials, Carrollton, Texas
  - Victorium Clinical Research, Houston, Texas
  - Southern Star Research Institute, LLC, San Antonio, Texas
- Argentina (3):
  - GEDYT, AAI
  - Sanatorio Maipu, Maipú
  - HIGEA, Mendoza
- Australia (5):
  - Monash Medical Centre, Clayton
  - Concord Repatriation General Hospital, Concord
  - St Vincents Hospital Melbourne, Fitzroy
  - John Hunter Hospital, New Lambton Heights
  - Mater Hospital Brisbane, South Brisbane
- Universitair Ziekenhuis Leuven, Leuven, Belgium
- Brazil (3):
  - Hospital das Clinicas do HC/UFMG, Belo Horizonte
  - CDC - Centro Digestivo de Curitiba, Curitiba
  - Pesquisare Saude, Santo André
- Canada (6):
  - GIRI Gastrointestinal Research Institute, Vancouver, British Columbia
  - Viable Clinical Research, Kentville, Nova Scotia
  - Barrie GI Associates, Barrie, Ontario
  - London Digestive Disease Institute, London, Ontario
  - ABP Research Services Corp., Oakville, Ontario
  - Toronto Immune and Digestive Health Institute Inc, Toronto, Ontario
- China (14):
  - Capital Medical University, Beijing Friendship Hospital, Beijing
  - Changzhou No 2 Peoples Hospital, Changzhou
  - Chongqing General Hospital, Chongqing
  - The First People's Hospital of Foshan, Foshan
  - The First Affiliated Hospital Sun Yat sen University, Guangzhou
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Affiliated Hospital of Hainan Medical University, Haikou
  - Huizhou Central People's Hospital, Huizhou
  - Zhongda Hospital Southeast University, Nanjing
  - Ningbo medical center lihuili hospital, Ningbo
  - Second Affiliated Hospital of Soochow University, Suzhou
  - The 2nd Affiliated Hospital & Yuying Children s Hospital Wenzhou Medical University, Wenzhou
  - Northern Jiangsu Peoples Hospital, Yangzhou
  - ZhuZhou Central Hospital, Zhuzhou
- Czechia (7):
  - Vojenska nemocnice Brno, Brno
  - Centrum gastroenterologie a hepatologie s.r.o., Kladno
  - PreventaMed, s.r.o., Olomouc
  - Gastromedic, Ltd., Pardubice
  - AXON Clinical s.r.o., Prague
  - Clinoxus s r o, Prague
  - MUDr. Michal Konecny, Ph.D. s.r.o., Přerov
- France (12):
  - CHU de Clermont Ferrand - Site Estaing, Clermont-Ferrand
  - APHP - Hopital Henri Mondor, Créteil
  - Institut Prive MICI Clinique des Cedres, Échirolles
  - CHU de Lille Hopital Claude Huriez, Lille
  - CHU de Montpellier Hopital Saint Eloi, Montpellier
  - Jules Verne Clinic, Nantes
  - CHU de Nice Hopital de l Archet, Nice
  - Hopital Saint-Antoine, Paris
  - Hospices Civils de Lyon CHU Lyon Sud, Pierre-Bénite
  - CHU Saint Etienne Hopital Nord, Saint-Priest-en-Jarez
  - CHU Toulouse - Hopital de Rangueil, Toulouse
  - CHRU de Nancy - Hopitaux de Brabois, Vandœuvre-lès-Nancy
- Germany (4):
  - Medizinisches Versorgungszentrum (MVZ) Dachau, Dachau
  - Praxisgemeinschaft Jerichow, Jerichow
  - Eugastro GmbH, Leipzig
  - Universitaetsmedizin Rostock, Rostock
- Greece (3):
  - Evangelismos S A, Athens
  - University General Hospital of Heraklion, Heraklion
  - Ippokratio General Hospital Of Thessaloniki, Thessaloniki
- Hungary (2):
  - Semmelweis Egyetem, Budapest
  - Pannónia Magánorvosi Centrum Kft, Budapest
- Israel (10):
  - Ha'Emek Medical Center, Afula
  - Assuta MC, Ashdod
  - Shamir Medical Center Assaf Harofeh, Be’er Ya‘aqov
  - Bnai Zion Medical Center, Haifa
  - Rambam Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Galilee Medical Center, Nahariya
  - Rabin Medical Center, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Istituto Clinico Humanitas, Rozzano, Italy
- Japan (24):
  - Juntendo University Hospital Urayasu, Chiba
  - Fukui Prefectural Hospital, Fukui-shi
  - Gamagori City Hospital, Gamagōri
  - National Hospital Organization Mito Medical Center, Higashiibaraki-gun
  - Kagoshima IBD Gastroenterology Clinic, Kagoshima
  - Tsujinaka Hospital Kashiwanoha, Kashiwa
  - Hospital of the University of Occupational and Enviromental Health, Kitakyushu
  - Japanese Red Cross Kumamoto Hospital, Kumamoto
  - Takano Hospital, Kumamoto
  - Kyorin University Hospital, Mitaka
  - Takagi Clinic, Miyagi
  - Hyogo Medical University Hospital, Nishinomiya Shi
  - Nakagami Hospital, Okinawa
  - Kinshukai Infusion Clinic, Osaka
  - National Hospital Organization Osaka National Hospital, Osaka
  - Osaka Metropolitan University Hospital, Osaka
  - Saga University Hospital, Saga
  - Toho University Sakura Medical Center, Sakura
  - Sapporo Tokushukai Hospital, Sapporo
  - Hokkaido P.W.F.A.C. Sapporo-Kosei General Hospital, Sapporo
  - Sapporo IBD Clinic, Sapporo
  - Tokyo Yamate Medical Center, Shinjuku-ku
  - Matsuda Hospital, Shizuoka
  - National Hospital Organization Shizuoka Medical Center, Sunto-gun
- Malaysia (6):
  - Hospital Sultanah Bahiyah, Alor Star
  - Hospital Ampang, Ampang
  - Hospital Sultanah Aminah, Johor Bahru
  - Hospital Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Tuanku Jaafar, Seremban
- Poland (12):
  - Centrum Medyczne Medis, Bydgoszcz
  - NZOZ Centrum Medyczne KERmed, Bydgoszcz
  - Centrum Medyczne Plejady, Krakow
  - Medrise Sp. z o.o., Lublin
  - RiverMED, Poznan
  - Endoskopia Sp z o.o., Sopot
  - Twoja Przychodnia - Szczecinskie Centrum Medyczne, Szczecin
  - Sonomed Sp. z o.o., Szczecin
  - GASTROMED Sp. z o.o., Torun
  - Bodyclinic Sp. z o.o. sp. k, Warsaw
  - Medical Network WIP Warsaw IBD Point Profesor Kierkus, Warsaw
  - Centrum Medyczne Oporow, Wroclaw
- Portugal (2):
  - Uls Braga - Hosp. Braga, Braga
  - Uls Loures Odivelas - Hosp. Loures, Loures
- Romania (2):
  - S C Delta Health Care S R L, Bucharest
  - Spitalul Clinic Colentina, Bucharest
- Spain (4):
  - Hosp. Clinic de Barcelona, Barcelona
  - Hosp. Univ. Infanta Leonor, Madrid
  - Hosp. Virgen Macarena, Seville
  - Hosp. Univ. I Politecni La Fe, Valencia
- Sweden (3):
  - Ersta sjukhus, Stockholm
  - Karolinska Universitetssjukhuset Solna, Stockholm
  - Akademiska Sjukhuset, Uppsala
- Taiwan (5):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District
- Turkey (Türkiye) (7):
  - Hacettepe University Hospital, Ankara
  - Gazi University Hospital, Ankara
  - Koc University, School of Medicine, Koc University Hospital, Istanbul
  - Ege Universitesi Tip Fakultesi, Izmir
  - Izmir Sehir Hastanesi, Izmir
  - Kocaeli University Medical Faculty, Kocaeli
  - Mersin University Medical Faculty, Mersin
- United Kingdom (8):
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - Glasgow Royal Infirmary, Glasgow
  - Fairfield General Hospital, Greater Manchester
  - Whipps Cross University Hospital, London
  - Guy's Hospital, London
  - St Georges University Hospital NHS Foundation Trust, London
  - Whiston Hospital, Rainhill
  - Stepping Hill Hospital, Stockport

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency